CLINICAL TRIAL: NCT05757453
Title: BoostOne Study (MHealth)
Brief Title: Boost Study 31380 (mHealth)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NXTech (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NX-31380; 1R43DA051270 (NIH)
Record Dates: First submitted 2023-01-31; First posted 2023-03-07 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Addiction
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental (Experimental): mHealth group
  Interventions: Device: mHealth

INTERVENTIONS:
Device: mHealth — Mobile platform

SUMMARY:
The purpose of this research is to examine the potential for a new software-based behavioral support approach, for individuals with opioid use disorder, as an addition to usual care.

DETAILED DESCRIPTION:
The purpose of this study is to examine the potential for a novel computer-based approach to mitigate the symptoms of opioid use disorder as part of a comprehensive treatment program. The study is designed as a single-arm field-test of cognitive training for individuals under supervised medical treatment for opioid use disorder. A custom and proprietary smartphone package (mHealth platform) comprises the intervention available to enrolled subjects for interaction over the study period. Commercial mobile devices serve as information presentation and data recording instruments. Additional outcome measures incorporate subject-reported data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Diagnosis of opioid use disorder
* Experiencing symptoms multiple times per week
* Familiar with smartphone usage

Exclusion Criteria:

- None specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Vien, MD, Principal Investigator — PHNY
Locations (1):
- PHNY, Astoria, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: MHealth group
  MHealth: Mobile application
Period: Overall Study
Arm/Group | Experimental
Started | 43
Completed | 21
Not Completed | 22

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 14
  Male | 29
  Declined to Report | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 15
  More than one race | 2
  Unknown or Not Reported | 22

OUTCOME MEASURES:

1. Primary Outcome: Interaction Engagement, as Assessed by Interactions Completed
Description: Interactions Completed (interactions completed, range 0 to unbound)
Time Frame: At 8 weeks
Measure: Mean (Full Range); unit: interactions
Arm/Group | Experimental
Number analyzed (Participants) | 43
interactions | 7.3 [1 to 28]

2. Secondary Outcome: Intervention Usability Rating, as Assessed by Likert User Experience Scale
Description: Subjective scoring of design and function usability, Likert User Experience Scale (score range 1-5, higher better)
Time Frame: At 8 weeks
Population: 18 of 21 participants did not complete survey at 8 week outcome measure time frame, resulting from technical error in survey delivery. 3 participants were analyzed.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 3
units on a scale | 4.7 [4 to 5]

3. Secondary Outcome: Treatment Progress Measure, as Assessed by TEA Score
Description: Patient-Centered instrument for evaluating progress, TEA Score (scale range 4 to 40, higher better), assessed weekly for 8 weeks with week 8 reported
Time Frame: At 8 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 21
score on a scale | 19 [15 to 36]

ADVERSE EVENTS:
Time Frame: 2 months, up to 3 months
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT05757453/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT05757453/SAP_001.pdf